CLINICAL TRIAL: NCT03734432
Title: IGAR-Breast Teleoperative Clinical Investigation
Brief Title: IGAR-Breast TeleOp Trial
Acronym: IGAR-Breast-TO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IGAR-TO-007
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer
Keywords: Diagnostic, Imaging, MRI
MeSH Terms: conditions — Breast Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): IGAR-Breast TeleOp
  Interventions: Device: IGAR-Breast TeleOp

INTERVENTIONS:
Device: IGAR-Breast TeleOp — Upon consent, each participant will undergo a teleoperative breast biopsy at their local site using the IGAR-Breast system, while the radiologist operates the system from a remote site.

SUMMARY:
The aim of this study is to answer the question: can the IGAR-Breast safely and effectively perform teleoperative breast biopsies? This is a prospective, pilot trial. 5-10 participants will be selected by the radiologist and the success of biopsy analyzed. In addition the number of adverse events, device events and procedural deviations will be assessed to determine safety and efficacy.

DETAILED DESCRIPTION:
In this prospective clinical trial, patients who present to the breast cancer clinic at one of the primary sites with suspected breast cancer requiring MRI-guided biopsy for diagnosis or staging will be screened consecutively. Patients who meet the inclusion criteria will be approached for consent to participate in the study. Upon consent, each participant will undergo a teleoperative breast biopsy at their local site using the IGAR-Breast system, while the radiologist operates the system from a remote site. All consenting participants will be followed up for the assessment of the secondary outcome measure.

A total of 5-10 participants will be consented for the pilot investigation.

Each individual subject's participation is estimated to last approximately one week post procedure, with the trial itself expected to be completed within one year of its start date.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged ≥ 18 years who require MRI-guided breast biopsy for diagnosis and/or staging Subjects are able to tolerate procedures for the MRI

Exclusion Criteria:

* Subjects who refuse or are unable to give free and informed consent Subjects requiring more than one breast biopsy Subjects with breast implants or other foreign bodies Subjects for whom investigator determines IGAR-Breast enabled MRI-guided breast biopsy is not possible (size of subject, location of lesion, size of breast, etc.) Subjects who are pregnant or who plan to become pregnant during the course of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects aged ≥ 18 years who require MRI-guided breast biopsy for diagnosis and/or staging Subjects are able to tolerate procedures for the MRI
Enrollment: 10 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
ability for IGAR-Breast to perform breast biopsies teleoperatively | at time of sampling and pathological evaluation
  analyzing the frequency of successful biopsy, in which the samples collected are of diagnostic quality as determined by radiologist

SECONDARY OUTCOMES:
number and frequency of adverse events, device events and procedural deviations in addition to a comparison to results from previous trials for efficacy | During procedure
  The number of times the local radiologist is required to participate will also be observed from a safety perspective

CONTACTS AND LOCATIONS:
Overall Officials: Mehran Anvari, Principal Investigator — Csii/St Joseph's Healthcare Hamilton
Locations (3):
- Canada (3):
  - St. Josephs Healthcare Hamilton, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Imagix - Radiologie Saint-Laurent, Saint-Laurent, Quebec

IPD SHARING:
Plan to Share IPD: No